CLINICAL TRIAL: NCT06805513
Title: Actual Use Trial to Switch Tadalafil 5 mg Tablets From Prescription to Over-the-Counter
Brief Title: Actual Use Trial of Tadalafil 5 mg
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUT16661; AUT16661 (Other: Sanofi Identifier); U1111-1267-2510 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-01-17; First posted 2025-02-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cialis OTC (Other): Open Label Single Arm study in men who have the symptoms of ED and who have an interest in an OTC treatment.
  Interventions: Combination Product: Tadalafil 5 mg tablets with a digital tool.

INTERVENTIONS:
Combination Product: Tadalafil 5 mg tablets with a digital tool. — The combination product will be a Drug (Tadalafil 5 mg) and Health Survey Assessment (as a mandatory digital tool). Tadalafil 5 mg will be taken orally, 1 tablet daily to use for treatment of erectile dysfunction. This study will be conducted remotely, via video interaction.
  Other Names: Cialis 5 mg

SUMMARY:
The purpose of this actual use trial (AUT) is to evaluate if participants can appropriately select and use the study product [Cialis over the counter (OTC)] using the labeling and the mandatory health survey assessment (HSA) for duration of 4-months.

DETAILED DESCRIPTION:
This will be an open-label 4-month AUT of tadalafil 5 mg tablet in men who are interested in an OTC treatment for erectile dysfunction. The open-label study will enroll approximately 2,250 participants who qualify for treatment based on the data they enter into the HSA of which an estimated 1000 participants will ultimately proceed to the use phase.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in Part II (enrolment phase) if they are:

1. Male or female, 16 years of age or older
2. Living in the US (Since this study will be conducted remotely, it is important to assure that all participants reside in this country.)

Participants will be included in Part III (use phase) if they:

1. Are male (sex assigned at birth)
2. Are at least 18 years of age
3. Complete the HSA with a purchase code for Cialis OTC
4. Purchase the study product

Exclusion Criteria:

Below participants will be excluded from Part II:

1. Participant lives in the state of Massachusetts (Massachusetts state law requires an application to the State Board of Pharmacy in order to get authorization to distribute the study product to participants who live there.)
2. Participant 18 years of age or older is unable or unwilling to show a current government-issued identification (ID) in order to verify identity and age
3. Participant cannot read, speak, and understand English
4. Participant has participated in another health-related market research study, product label study, or clinical trial in the past 12 months
5. Participant has ever participated in a research study about a medicine for erectile dysfunction
6. Participant, or someone else in the household works for a pharmaceutical company
7. Participant, or someone else in the household is a healthcare professional, works as a part of a health care practice, or has been trained as a healthcare professional
8. Participant, or someone else in the household is employed by a market research or advertising company
9. Participant or someone else in the household is employed by PEGUS Research
10. Participants will be told that if they need corrective lenses to read, they must have them when the remote Enrollment Interview is conducted (Part II). If they do not, they will not be allowed to participate. This exclusion will be implemented during the remote Subgroup Identification Interview (SGI) Interview where the participants will be re-screened.
11. Participants who are considered minors, according to the law in the state where they reside, who do not have a parent or guardian present and willing to electronically sign permission to allow the minor to participate in the SGI and Enrollment Interviews. A participant is considered a minor in all states if they are 16-17 years of age. Additionally, participants 18 years of age in Alabama or Nebraska, and participants 18-20 years of age in Mississippi are also considered minors.
12. Participant is not willing or able to attend/participate in the Enrollment Interview remotely
13. Participant, or someone else in the household, has participated in this study (only one member of each household will be allowed to participate)
14. Participant does not provide verbal permission to video record study interviews
15. If necessary to obtain approximately 30% low health literacy (LHL), participants who are not LHL will be screened out

Below participants will be excluded from Part III:

1. Participants who were not excluded for DNU conditions in the HSA, but were determined in the Medical Assessment to have any of the DNU conditions listed on the DFL
2. Participants who do not sign the Informed Consent Document (ICD) or if the parent or guardian of a minor does not sign the ICD. (Parent/guardian refusal applies to males who are 18 years of age or older but considered minors in the state where they reside.)
3. Participants who are unwilling to provide contact information
4. Participants who are unwilling or unable to use an eDiary to record the required information
5. Participants who the principal investigator or the Medical Monitor believes should be excluded or removed from further participation in the Use Phase due to safety concerns

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 2250 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of inter-dosing intervals in which the recommended time between doses is followed | From the beginning of Use phase to end, at 120 days.
  Dosing intervals from participant dosing occasions as recorded in the eDiary population will be used to calculate this endpoint.
The proportion of all participants found to have a do not use (DNU) condition in the Medical Assessment who also received a DNU Outcome screen in the Health survey assessment | 1 day (completion of the enrollment interview)

SECONDARY OUTCOMES:
Descriptive analysis of care-seeking behaviors in the case of heart attack, priapism, allergic reaction, sudden vision or hearing loss, where the participant took Cialis OTC within the 72 hour time period prior to the event | From the beginning of Use phase to end, at 120 days.
Descriptive analysis of care-seeking behaviors associated with dizziness or feeling faint which does not get better after sitting or lying down, and where the participant took Cialis OTC within the 72 hour time period prior to the event | From the beginning of Use phase to end, at 120 days.
Descriptive analysis of serious adverse event (SAE)s and adverse event of special interest (AESI)s. | From the beginning of Use phase to end, at 150 days (120 days study period + 30 day follow-up period).
Descriptive analysis of dosing behavior patterns among those who do not comply with the recommended dosing interval. | From the beginning of Use phase to end, at 120 days.
The proportion of participants ever prescribed a nitrate medicine who also received a DNU-Nitrate Outcome screen in the HSA. | 1 day (completion of the enrollment interview)
The proportion of all participants found to have ask a doctor before use (AADBU) or ask a doctor or pharmacist before use (AADPBU) conditions in the Medical Assessment who also received an AADBU or AADPBU Outcome screen in the HSA. | 1 day (completion of the enrollment interview)
The proportion of participants who take 1 tablet (5 mg) on the first dosing occasion. | From the beginning of Use phase to end, at 120 days.
The proportion of dosing occasions in which 2 tablets (10 mg) are not exceeded per dosing occasion. | From the beginning of Use phase to end, at 120 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Pegus, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org